CLINICAL TRIAL: NCT02128438
Title: Most People With Low Back Pain Have Associated Cervicothoracic Musculoskeletal Dysfunction: an Observational Study
Status: Completed | Type: Observational
Sponsor: Swami Vivekanand National Institute of Rehabilitation Training and Research (Other)
Responsible Party: Principal Investigator, P.P.Mohanty, Associate Professor in Physiotherapy, Swami Vivekanand National Institute of Rehabilitation Training and Research
Other Study IDs: mohanty0202
Record Dates: First submitted 2014-04-25; First posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In general , the diagnosis of back pain can be broken into three major categories: Mechanical ( Osteoarthritis , Spinal stenosis , Spondylolisthesis) ; Non- mechanical ( Tumor , Infection , Inflammatory arthritis ) and Miscellaneous (Osteoporosis , Psychosomatic disorders , neuropathic joints , visceral diseases ). Although 98% of LBP may be caused by mechanical factors, it is the other 2% caused by malignancy, infection, visceral diseases and other red herrings that must be considered most seriously.

The investigators have observed in their practice that lateral pressure on 5th lumbar vertebra sometimes gives rise to cervicothoracic pain and central PA pressure over cervicothoracic spines reproduce original low back and leg pain. So the question arises whether Cervico-thoracic dysfunction is associated with low back pain with or without radiation to lower extremities?

ELIGIBILITY:
Inclusion Criteria:

* mechanical low back pain with or without radiation to lower limb.

Exclusion Criteria:

* any recent trauma or fractures to cervico-thoracic junction, osteoporosis, inflammatory arthritis, tuberculosis, bone disease, congenital deformity
* vascular disorders
* rapidly progressing neurological deficits
* sudden onset of neurological deficits and all red flags to manual therapy.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Persons with low back pain who had attended our hospital and sub centres with a complaint of low back pain
Sampling Method: Non-Probability Sample
Enrollment: 940 (Actual)
Dates: Start 2007-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
incidence of cervico-thoracic dysfunction in patients with low back pain | The outcome measure, viz. the incidence of cervico-thoracic dysfunction was ascertained immediately at the time of initial physical assessment. No follow-up was required.
  incidence of cervico-thoracic dysfunction in patients with low back pain with or without radiation down the lower extremity, which is characterized by reproduction of the original symptom by central PA pressure of cervicothoracic spines and digital pressure by algometer over levator scapulae

CONTACTS AND LOCATIONS:
Overall Officials: Patitapaban Mohanty, PhD, Principal Investigator — Swami Vivekanand National Institute of Rehabilitation Training and Research; Basant K Behera, M.S (Ortho), Study Chair — SCB medical college and hospital, Cuttack
Locations (1):
- SVNIRTAR, Olatpur, Cuttack Dt, Odisha, India